CLINICAL TRIAL: NCT03610529
Title: CardioSenseSystem Compared to Philips Telemetry System Regarding Efficacy and Safety in the Monitoring of ECG
Brief Title: CardioSenseSystem Compared Study Regarding Efficacy and Safety in the Monitoring of ECG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Novosense AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NovoECG; 5.1-2018-18343 (Registry Identifier: Swedish Medical Products Agency); 2018/9 (Registry Identifier: Regional Ethical Review Board in Lund, Sweden)
Record Dates: First submitted 2018-07-23; First posted 2018-08-01 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Cardiac Arrythmias; Unstable Angina; Heart Valve Disorders; Disorder of Aorta
Keywords: ECG Monitoring; Controlled; Comparative; Clinical trial
MeSH Terms: conditions — Angina, Unstable; Heart Valve Diseases; Aortic Diseases

STUDY DESIGN:
Intervention Model Description: The study participants will be using both the experimental device and the control device simultaneously throughout the study participation. The participant will thereby act as its own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ECG monitoring system CardioSenseSystem group (Experimental)
  Interventions: Device: CardioSenseSystem
- ECG monitoring system Philips Intellivue (Active Comparator)
  Interventions: Device: Philips Intellivue

INTERVENTIONS:
Device: CardioSenseSystem — CardioSensySystem is a novel wireless ECG monitoring system developed by Novosense AB for monitoring of ECG in health care departments.
  Arms: ECG monitoring system CardioSenseSystem group
Device: Philips Intellivue — Philips Intellivue in an established ECG monitoring system used at the clinical investigational device.
  Arms: ECG monitoring system Philips Intellivue

SUMMARY:
This is a prospective, controlled, comparative clinical trial of a new ECG monitoring system CardioSenseSystem prior CE marking. The aim of the study is to demonstrate that the CardioSenseSystem's cable-free ECG monitoring system (investigational device) is equivalent or better than traditional and accepted industry standard for cable-based ECG monitoring system (control device). In this study accepted industry standard is Philips Intellivue. In order to investigate this, the study will measure ECG monitoring interruptions, management time and alarm performance. The study population will consist of sixty (60) adult subjects requiring ECG and that are fulfilling the eligibility criteria for study participation. The subjects will be using both the investigational device and the control device simultaneous for measuring data loss, management time and alarm function up to 24 hours.

DETAILED DESCRIPTION:
A prospective, controlled and comparative clinical trial before CE marking of a new ECG monitoring system CardioSenseSystem. The study population will consist of sixty (60) adult subjects requiring ECG and that are fulfilling the eligibility criteria for study participation. The subjects will be monitored by both the investigational device and the control device for measuring data loss, management time and alarm function up to 24 hours. The duration of the study is estimated to 4 months.

CardioSenseSystem is designed to provide wireless high-quality ECG monitoring. The system developed by Novosense AB consists of three components: the CardioPatch, the Novosense Base Station and the Back-End System. The CardioPatch is a wireless sensor capable to record and transmit ECG data. The CardioPatch send ECG data to the Novosense Base Station, which is the receiving unit. The Back-End System is used for presentation, storage and processing of ECG information. The CardioPatch sensor is applied to the body with an adhesive in the same way as a traditional ECG electrode. In contrast, the CardioPatch is a fully integrated unit containing electrodes, ECG amplifier and a radio transmitter. Novosense's wireless ECG sensors, CardioPatch, transmits the ECG signal 24 hours to the Novosense Base Station receiver.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years old.
2. Patient hospitalized at the investigational site and in need of ECG monitoring.
3. Patient with expected alarms during the 24 hours ECG monitoring.
4. Patient who has been informed of the clinical trials purpose, limitations and relevance, and who has voluntarily agreed to participation in the clinical trial by signing the informed consent form.

Exclusion Criteria:

1. Patient with burns.
2. Patient with known allergy or sensitivity to any of the compositions in CardioPatch.
3. Patient with infection in the area where the electrodes are to be placed.
4. Patient with fragile skin (eg after prolonged cortisone treatment).
5. Patient with open sternum / sternum (eg severe heart failure postoperatively) or treatment for infection of the sternum.
6. Patient with mechanical auxiliary heart or ECMO.
7. Patient with implantable defibrillator.
8. Severely ill patient during end of life.
9. Patient participating in any other clinical trial.
10. Patient where the investigator judge that participation may be risky for the patient or obstruct or interfere the implementation of the trial as approved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Lost of monitoring data | During 24 hour per subject
  Compare time of interruptions in the monitoring system between the investigational device and the control device.

SECONDARY OUTCOMES:
Management time | During 24 hour per subject
  Compare management time between the investigational device and the control device. This is done by measuring the time required for the sterilization of cables, battery replacements, application of electrodes and cables, and extra management time for applying electrodes and cables if unconnected.
Number of correct yellow and red alarm | During 24 hour per subject
  Compare the number of correct yellow and red alarm between the investigational device and the control device.
Number of false yellow and red alarm | During 24 hour per subject
  Compare the number of false yellow and red alarm for the investigational device and the control device.
Incidence and severity of Averse Events | During 24 hour per subject
  The incidence and severity of adverse events associated with the investigational device and the control device.

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Linnér, MD PhD EDIC, Principal Investigator — Skane University Hospital
Locations (1):
- VO Thorax o Kärl, Region Skåne, Lund, Entrégatan 7, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sponsors website — http://www.novosense.se